CLINICAL TRIAL: NCT03413696
Title: Effects of Health Literacy and Hepatitis C Knowledge on Hepatitis C Treatment Willingness in HIV-coinfected Patients, According to Hepatitis C Treatment Referral Status
Brief Title: Effects of Health Literacy and HCV Knowledge on HCV Treatment Willingness in HIV-coinfected Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward Cachay, MD, MAS, Associate Professor of Clinical Medicine, University of California, San Diego
Other Study IDs: 20170991; 170218 (Other: UCSD Human Research Protections Program)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C; Hepatitis C, Chronic; HIV/AIDS
Keywords: HIV; Health literacy; Hepatitis C; Hepatitis C knowledge; HIV knowledge; Hepatitis C treatment
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Not referred for HCV therapy
- Referred for HCV therapy,did not show up
- Referred,attended HCV therapy evaluation

SUMMARY:
A clinical observational study for patients with HIV co-infected with hepatitis C that investigates the levels of their health literacy, hepatitis C and HIV knowledge. Participants will complete a one-time assessment of these studied domains and categorized in three groups defined by their hepatitis C treatment referral status: not-referred, referred-attended, referred and no-show.

DETAILED DESCRIPTION:
The main purpose of this research study is to investigate the prevalence of inadequate health literacy and hepatitis C knowledge and their determinants among people living with HIV/AIDS co-infected with hepatitis C. The observation will determine if health literacy and/or hepatitis C knowledge are predictors of patient willingness and intention to be treated for HCV in the overall cohort and stratified according to study groups as noted above.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥ 18 years) HIV-infected patient attending the UCSD Owen Clinic
* Regardless of ethnic background
* English or Spanish speaking
* With active HCV infection defined as having a detectable HCV viral load with or without a positive HCV antibody

Exclusion Criteria:

* Neurocognitive impairment precluding participation
* Physical illness precluding participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living with HIV, coinfected with HCV, who are receiving care at the UCSD Owen Clinic at the time of data collection
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Inadequate health literacy (s-TOFHLA inventory) | Baseline before HCV treatment consideration
  The primary outcome will measure the point prevalence of inadequate health literacy among persons with HIV/AIDS with active hepatitis C infection.

SECONDARY OUTCOMES:
Hepatitis C knowledge (using the modified Treolar's scale) | Baseline before HCV treatment consideration

OTHER OUTCOMES:
Determinants of inadequate health literacy and HCV knowledge | Baseline before HCV treatment consideration
  To ascertain determinants of inadequate health literacy and HCV knowledge among PLWH coinfected with HCV in the overall study group and stratified according to group membership: (1) not referred for HCV therapy, (2) those referred but no show, and (3) those referred and attended HCV therapy.
Predictors of patient willingness to HCV treatment | Baseline before HCV treatment consideration
  To ascertain predictors of patient willingness and intention to be treated for HCV with particular attention to the independent effect of health literacy and HCV knowledge in the overall cohort and stratified according to study groups as noted above.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Cachay, MD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- Owen Clinic - University of California, San Diego, San Diego, California, United States